CLINICAL TRIAL: NCT01831024
Title: Clinical Performance, Efficacy and Safety of the DigniCap™ System, a Scalp Hypothermia System, in Preventing Chemotherapy Induced Alopecia in Patients With Early Stage Breast Cancer
Brief Title: Efficacy and Safety of Dignicap System for Preventing Chemotherapy Induced Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Target Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DIG-001
Record Dates: First submitted 2013-04-03; First posted 2013-04-15 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Chemotherapy Adjuvant; Breast Cancer
Keywords: Cold cap; Scalp cooling; Chemotherapy induced alopecia; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Dignicap System
  Interventions: Device: Dignicap System
- Control Group (No Intervention): Concurrent age and chemotherapy matched control

INTERVENTIONS:
Device: Dignicap System — The DigniCap™ System consists of the digitized system for controlled scalp cooling (Digni C3) in conjunction with the soft, tight-fitting silicon cap (DigniCap™), the neoprene outer cap (DigniTherm™), and the liquid coolant (DigniCool). DIGNISTICK™ is prepared to log data from a treatment when inserted in the slot. DIGNICARD™ is a key card which has to be inserted in order to start a treatment.
  Other Names: Cold cap
  Arms: Treatment Group

SUMMARY:
The efficacy and safety of the Dignicap System to prevent chemotherapy induced alopecia will be evaluated in women with early breast cancer undergoing adjuvant or neoadjuvant chemotherapy regimens. The scalp cold cap will be applied at each chemotherapy cycle. Hair loss will be evaluated by patient self assessment of 5 standardized photographs taken prior to each chemotherapy cycle. A concurrent control group not using a cold cap will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female patients >/= 18 years of age
* Documented diagnosis of stage I or II breast cancer
* A planned course of chemotherapy in the adjuvant or neoadjuvant setting with curative intent including one of the following regimens:

  * Doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 x 4 - 6 cycles IV every 2 - 3 weeks
  * Docetaxel 75 mg/m2 and cyclophosphamide 600 mg/m2 x 4 - 6 cycles IV every 3 weeks
  * Paclitaxel 80 mg/m2 weekly IV x at least 12 weeks with or without IV trastuzumab
  * Paclitaxel 175 mg/m2 IV every 2 weeks x 4 - 6 cycles (without an anthracycline)
  * Paclitaxel weekly and carboplatin AUC 2 weekly or AUC 6 every 3 weeks IV x 4 - 6 cycles and trastuzumab IV weekly or every 3 weeks
  * Docetaxel 75 mg/m2 and carboplatin AUC 6 IV every 3 weeks x 4 - 6 cycles and trastuzumab IV weekly or every 3 weeks
  * Targeted agents such as trastuzumab or lapatinib are allowed
* Plan to complete chemotherapy within 6 months
* At least two years out from the last chemotherapy causing hair loss with complete recovery of hair
* Karnofsky performance status >/= 80%
* Willing and able to sign informed consent for protocol treatment
* Willing to participate in study procedures including having photographs of the head before the first cycle of chemotherapy and 1 month after the last chemotherapy
* Willing to enroll in an extension protocol for follow up for 5 years following the end of chemotherapy treatment

Exclusion Criteria:

* Patients with female pattern baldness resembling picture I-3 or higher on the Savin scale
* Autoimmune disease affecting hair; e.g. alopecia areata, systemic lupus with associated hair loss
* A history of whole brain radiation
* Plans to use a chemotherapy regimen other than those specified in the inclusion criteria. Specifically, patients receiving a regimen including both an anthracycline and a taxane are not eligible for this trial (AC/T, EC/T, TAC, etc.)
* Concurrent hormone therapy with chemotherapy. Hormone therapy should be used as indicated following completion of chemotherapy
* Underlying clinically significant liver disease including active viral hepatitis with abnormal liver function tests >1.5 times the upper limit of normal, including alkaline phosphatase, AST, and total bilirubin. Patients with Gilbert´s disease (elevated indirect bilirubin only) will be eligible for participation.
* Clinically significant renal dysfunction defined as serum creatinine > upper limit of normal.
* A serious concurrent infection or medical illness which would jeopardize the ability of the patient to complete the planned therapy and follow-up
* A history of persistent grade 2 (or higher) alopecia induced by prior chemotherapeutic regimens
* Participation in any other clinical investigation or exposure to other investigational agents, drugs, device or procedure that may cause hair loss
* Intercurrent life-threatening malignancy
* A history of cold agglutinin disease or cryoglobulinemia.
* Evidence of untreated or poorly controlled hyper or hypothyroidism
* A history of silicon allergy
* American Society of Anesthesiologist Class ≥3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-07; Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hair loss | 4 weeks after last chemotherapy cycle
  5 standardized photographs will be evaluated by the patient using the Dean Scale for alopecia

SECONDARY OUTCOMES:
Tolerability | Every 2 to 4 weeks for up to 12 weeeks
  The percentage of patients who complete all planned cycles of chemotherapy do so using the DigniCap™ System
Adverse events | 6 months
  spontaneous reporting by the patient or identified during physical examination
Hair regrowth | 4 Weeks after last chemotherapy
  Patient assessment using hair regrowth survey
Quality of Life | 4 Weeks after last chemotherapy cycle
  European Organization for Research and Treatment of Cancer-Quality of Life-BR23 questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Beth Israel Medical Center, Comprehensive Cancer Center, New York, New York
  - Weill Cornell Breast Center, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Rugo HS, Klein P, Melin SA, Hurvitz SA, Melisko ME, Moore A, Park G, Mitchel J, Bageman E, D'Agostino RB Jr, Ver Hoeve ES, Esserman L, Cigler T. Association Between Use of a Scalp Cooling Device and Alopecia After Chemotherapy for Breast Cancer. JAMA. 2017 Feb 14;317(6):606-614. doi: 10.1001/jama.2016.21038. PMID 28196257